CLINICAL TRIAL: NCT01891292
Title: A Phase 2 Study of the Efficacy of Antioxidant Therapy Compared With Enalapril in Slowing the Progression of Sickle Nephropathy in Children
Brief Title: Efficacy of Antioxidant Therapy Compared With Enalapril in Sickle Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of The West Indies (Other)
Collaborators: Caribbean Health Research Council (Other)
Responsible Party: Principal Investigator, Marvin Reid, Professor, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECP 172, 10/11
Record Dates: First submitted 2013-01-22; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Microalbuminuria; Sickle Cell Nephropathy
MeSH Terms: interventions — Enalapril; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention)
- Enalapril (Active Comparator)
  Interventions: Drug: Enalapril
- N-Acetylcysteine (Active Comparator)
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: Enalapril — 0.25-0.35 mg/kg/day
  Arms: Enalapril
Drug: N-Acetylcysteine — N-Acetylcysteine 0.5 mmol/kg
  Arms: N-Acetylcysteine

SUMMARY:
The purpose of this study is to determine whether enalapril or antioxidant therapy (N-Acetylcysteine) is effective in reducing microalbuminuria in children with sickle cell disease and and its progression to sickle nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Homozygous S sickle cell disease
* Diagnosed by newborn screening
* determined to have persistent microalbuminuria
* satisfied criteria for microalbuminuria screening
* parental consent

Exclusion Criteria:

* Asymptomatic bacteriuria on screening urine cultures
* On Hydroxyurea therapy
* Pre-existing complications of SCD which would meet local criteria for HU therapy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
urinary albumin excretion rate | 12 months

SECONDARY OUTCOMES:
Glomerular filtration rate | 12 months
  Measurement of glomerular filtration rate by iohexol

CONTACTS AND LOCATIONS:
Locations (1):
- Sickle Cell Unit, Kingston, Jamaica

REFERENCES:
- [Derived] Sasongko TH, Nagalla S. Angiotensin-converting enzyme (ACE) inhibitors for proteinuria and microalbuminuria in people with sickle cell disease. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD009191. doi: 10.1002/14651858.CD009191.pub4. PMID 34932828